CLINICAL TRIAL: NCT02398370
Title: Evaluate the Safety and Feasibility of Injecting Placental Matrix-Derived Mesenchymal Stem Cells Into the Penis to Treat the Symptoms of Mild to Moderate Erectile Dysfunction
Brief Title: Evaluate the Safety and Feasibility of Injecting PMD-MSC Into the Penis to Treat the Symptoms of Mild to Moderate ED
Acronym: PMD-MSC-ED-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melissa Marchand (Other)
Responsible Party: Sponsor-Investigator, Melissa Marchand, M.D., Z Urology
Organization: Z Urology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMD-MSC-ED-01
Record Dates: First submitted 2015-03-09; First posted 2015-03-25 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Erectile Dysfunction
Keywords: ED
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Injection of PMD-MSCs into the penis (Experimental): Subjects will receive an initial injection of 1.0cc of Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs). Subjects will be eligible for re-injection at 3 months and/or 6 months as determined by the clinician based patient reported treatment satisfaction.
  Interventions: Biological: Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs)

INTERVENTIONS:
Biological: Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs)
  Other Names: Ovation

SUMMARY:
Prospective, open-label, non-randomized, study to be conducted at a single center. Ten subjects will undergo an injection of Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs) into the penis for the treatment of mild to moderate erectile dysfunction. Follow up visits will be conducted at 6 weeks, 3 months, 6 months, and 12 months. Subjects will be evaluated for re-injection beginning at 3 months. Eligibility is determined by the clinician based on patient reported treatment satisfaction.

DETAILED DESCRIPTION:
An estimated 18 million men in the United States are diagnosed with Erectile Dysfunction (ED). ED is a physical condition triggered by a man's mental, emotional, and medical state. Defined by the repeated and consistent problem sustaining an erection suitable for sexual intercourse; ED can lead to performance anxiety and depression as a result partners of men with ED also suffer emotional and psychological effects.

Lifestyle, smoking, medical conditions such as diabetes, hypertension and vascular problems, prostate cancer and medication side effects all can contribute to the cause of ED.

Conservative treatments can begin with lifestyle change; natural remedies include the use of herbs such as L-Arginine, Ginko, Zinc, and Yohimbe. Prescription medications known as phosphodiesterase type 5 inhibitors are often used but are costly. other therapies involve the penis pump/penis vacuum, penile implants that offer a permanent solution and surgery to improve the blood flow to the penis can improve erections.

Mesenchymal stem cells (MSCs) have been used for a variety of medical treatments to repair and regenerate acute and chronically damaged tissues. These cells have the potential to repair human tissue by forming cells of mesenchymal origin, such as cartilage, bone, fat, muscle, and blood vessels. Most research has focused on bone marrow derived stem cells (BMC) however the process for harvesting the cells is invasive, painful, and yields a low cell count. The human placenta offers an alternative source form MSCs. Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs) are compromised of a novel cellular repair matrix derived from placental mesenchyme. Mesenchyme is the meshwork of embryonic connective tissue in the mesoderm, from which are formed the muscular and connective tissues of the body and also the blood vessels. PMD-MSCs provide the extracellular matrix viable mesenchymal stem cells (MSCs) that coordinate the tissue repair process, regenerative growth factors, and anti-inflammatory cytokines required to regenerate the damaged vasculature of the penile corpora.

Injecting PMD-MSCs into the penile corpora to replace the dysfunctional or dead cells is an intriguing option for cell-based treatment for ED. The research proposed here will establish the safety and feasibility of utilizing intracavernosal injections of PMD-MSCs to treat Erectile Dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 40-70
2. Willing and able to provide written informed consent
3. Chronic, organic erectile dysfunction (ED), duration at least 0.5 years, with baseline International Index of Erectile Function-Erectile Function (IIEF-EF) score greater than or equal to 21
4. Willing to complete questionnaires
5. Involved in a monogamous, heterosexual relationship for at least 3 months with both partners motivated to have or attempt sexual intercourse at least 4 times per month beginning two weeks after study treatment (subject reported)
6. Not interested or able to use oral PDE-5 inhibitor (PDE-5i) drug therapy, and willing to forgo these treatments for the first 6-month period following study treatment (in addition may include a 4-week washout since last PDE-5i use prior to completion of the baseline erectile function assessments and study treatment)
7. Willing to limit alcohol intake and eliminate use of recreational drugs for sexual encounters
8. Willing to undergo an injection 9 Mentally competent and able to understand all study requirements (based on investigator assessment)

10. Willing to be available for all baseline, treatment, and follow up examinations required by protocol 11. Willing to forego participation in any other study throughout the duration of this study

Exclusion Criteria:

1. Evidence of prostate cancer which requires additional radiotherapy or other adjuvant therapy
2. Previous pelvic or abdominal radiation therapy
3. Previous, concomitant or scheduled use of anti-androgen therapy
4. Untreated hypogonadism or low serum total testosterone (<200 ng/dL)
5. Clinically evident penile anatomical deformities (e.g., Peyronie's disease) or history of priapism
6. Skin irritation, infection, wound, sore, or disruption in the immediate areas of skin entry for penile injection
7. Use of any non-study treatment for erectile dysfunction within 4 weeks of study treatment and a lack of willingness to continue through 6 months after study treatment
8. Any previous penile implant or penile vascular surgery
9. Current or previous malignancy other than localized prostate cancer
10. Uncontrolled hypertension or hypotension (systolic blood pressure > 170 or <90 mm Hg, and diastolic blood pressure > 100 or < 50 mm Hg)
11. Reported unstable cardiovascular disease (e.g., unstable angina, myocardial infarction within the past 6 months, cardiac failure or life-threatening arrhythmia, congestive heart failure) or symptomatic postural hypotension within 6 months before screening
12. Current urinary tract or bladder infection
13. Drug, alcohol, or substance abuse reported within the last three years (subject reported) Subject's sexual partner < 18 years of age or has any gynecologic problems
14. Major medical conditions, or any other factors that would limit participation in sexual intercourse to less than 4 times per month (subject reported)
15. Weight less than 154lbs/ 70 kg, or BMI greater than or equal to 30
16. Systemic autoimmune disorder
17. Significant active systemic or localized infection
18. Receiving immunosuppressant medications

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Peak Systolic Velocity without trimix (cm/s) | Baseline
Peak Systolic Velocity without trimix (cm/s) | 6 weeks
Peak Systolic Velocity without trimix (cm/s) | 3 months
Peak Systolic Velocity without trimix (cm/s) | 6 months
Peak Systolic Velocity without trimix (cm/s) | 12 months

SECONDARY OUTCOMES:
End Diastolic Velocity without trimix (cm/s) | Baseline
End Diastolic Velocity without trimix (cm/s) | 6 weeks
End Diastolic Velocity without trimix (cm/s) | 3 months
End Diastolic Velocity without trimix (cm/s) | 6 months
End Diastolic Velocity without trimix (cm/s) | 12 months

OTHER OUTCOMES:
Peak Systolic Velocity with trimix (cm/s) | Baseline
Peak Systolic Velocity with trimix (cm/s) | 6 weeks
Peak Systolic Velocity with trimix (cm/s) | 3 months
Peak Systolic Velocity with trimix (cm/s) | 6 months
Peak Systolic Velocity with trimix (cm/s) | 12 months
End Diastolic Velocity with trimix (cm/s) | Baseline
End Diastolic Velocity with trimix (cm/s) | 6 weeks
End Diastolic Velocity with trimix (cm/s) | 3 months
End Diastolic Velocity with trimix (cm/s) | 6 months
End Diastolic Velocity with trimix (cm/s) | 12 months
Rigidity test (Pass / Fail) | Baseline
Rigidity test (Pass / Fail) | 6 weeks
Rigidity test (Pass / Fail) | 3 months
Rigidity test (Pass / Fail) | 6 months
Rigidity test (Pass / Fail) | 12 months
Stretched Penile Length before trimix (cm/s) | Baseline
Stretched Penile Length before trimix (cm/s) | 6 weeks
Stretched Penile Length before trimix (cm/s) | 3 months
Stretched Penile Length before trimix (cm/s) | 6 months
Stretched Penile Length before trimix (cm/s) | 12 months
Post Penile Width with trimix | Baseline
Post Penile Width with trimix | 6 weeks
Post Penile Width with trimix | 3 months
Post Penile Width with trimix | 6 months
Post Penile Width with trimix | 12 months
International Index of Erectile Function (IIEF) | Baseline
International Index of Erectile Function (IIEF) | 6 weeks
International Index of Erectile Function (IIEF) | 3 months
International Index of Erectile Function (IIEF) | 6 months
International Index of Erectile Function (IIEF) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Zahalsky, M.D., Principal Investigator — Z Urology
Locations (1):
- Z Urology, Coral Springs, Florida, United States

REFERENCES:
- [Derived] Levy JA, Marchand M, Iorio L, Cassini W, Zahalsky MP. Determining the Feasibility of Managing Erectile Dysfunction in Humans With Placental-Derived Stem Cells. J Am Osteopath Assoc. 2016 Jan;116(1):e1-5. doi: 10.7556/jaoa.2016.007. PMID 26745574